CLINICAL TRIAL: NCT04766086
Title: A PHASE 2B, PLACEBO-CONTROLLED, RANDOMIZED, OBSERVER-BLINDED TRIAL TO EVALUATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF A MULTIVALENT GROUP B STREPTOCOCCUS VACCINE WHEN ADMINISTERED CONCOMITANTLY WITH TETANUS, DIPHTHERIA, AND ACELLULAR PERTUSSIS VACCINE (TDAP) IN HEALTHY NONPREGNANT WOMEN 18 THROUGH 49 YEARS OF AGE
Brief Title: Trial to Evaluate the Safety, Tolerability, and Immunogenicity of A Multivalent Group B Streptococcus Vaccine When Administered Concomitantly With Tdap in Healthy Nonpregnant Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: C1091005
Record Dates: First submitted 2021-02-18; First posted 2021-02-23 (Actual); Results first posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-04

CONDITIONS: Group B Streptococcus Infections
MeSH Terms: interventions — Diphtheria-Tetanus-acellular Pertussis Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This is an observer-blinded study. Study staff dispensing and administering the vaccine will be unblinded, but all other study personnel, including the principal investigator, and the subject, will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- GBS6 and Tdap (Experimental): Multivalent group B streptococcus vaccine and Tetanus, diphtheria, and acellular pertussis vaccine (Tdap)
  Interventions: Biological: Multivalent Group B streptococcus vaccine; Biological: Tetanus, diphtheria, and acellular pertussis vaccine
- GBS6 and Placebo (Experimental): Multivalent group B streptococcus vaccine and Placebo
  Interventions: Biological: Multivalent Group B streptococcus vaccine; Biological: Placebo
- Placebo and Tdap (Experimental): Placebo and Tetanus, diphtheria, and acellular pertussis vaccine (Tdap)
  Interventions: Biological: Tetanus, diphtheria, and acellular pertussis vaccine; Biological: Placebo

INTERVENTIONS:
Biological: Multivalent Group B streptococcus vaccine — Multivalent Group B streptococcus vaccine
  Arms: GBS6 and Placebo; GBS6 and Tdap
Biological: Tetanus, diphtheria, and acellular pertussis vaccine — Tetanus, diphtheria, and acellular pertussis vaccine
  Other Names: Tdap
  Arms: GBS6 and Tdap; Placebo and Tdap
Biological: Placebo — Saline control
  Arms: GBS6 and Placebo; Placebo and Tdap

SUMMARY:
This phase 2B, placebo-controlled, randomized, observer-blinded trial will evaluate the safety, tolerability, and immunogenicity of the investigational multivalent group B streptococcus vaccine administered concomitantly with Tdap in healthy nonpregnant women 18 through 49 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women ≥18 and ≤49 years of age.
* Participants who are willing and able to comply with scheduled visits, investigational plan, laboratory tests, lifestyle considerations, and other study procedures, including completion of the e-diary from Day 1 to Day 7 following administration of investigational product.
* Healthy females at enrollment who are determined by medical history, physical examination, and clinical judgment of the investigator to be eligible for inclusion in the study.
* Expected to be available for the duration of the study and who can be contacted by telephone during study participation.
* Capable of giving personal signed informed consent.

Exclusion Criteria:

* Pregnant female participants; breastfeeding female participants; positive urine pregnancy test for women of childbearing potential (WOCBP) at Visit 1 (prior to vaccination)
* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the investigational product or any diphtheria toxoid-containing or CRM197-containing vaccine.
* History of microbiologically proven invasive disease caused by group B streptococcus.
* Immunocompromised participants with known or suspected immunodeficiency.
* Bleeding diathesis or condition associated with prolonged bleeding that would in the opinion of the investigator contraindicate intramuscular injection.
* Other acute or chronic medical or psychiatric condition, including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Previous vaccination with any licensed or investigational GBS vaccine, or planned receipt during the participant's participation in the study (through the 1-month follow-up visit [Visit 2]).
* Vaccination within 5 years with tetanus and diphtheria toxoids and acellular pertussis-containing vaccines (Tdap) before investigational product administration.
* Participants who receive treatment with immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids
* Vaccination with diphtheria- or CRM197-containing vaccine(s) from 6 months before investigational product administration, or planned receipt through the 1-month follow-up visit.
* Receipt or planned receipt of blood/plasma products or immunoglobulin, from 60 days before investigational product administration through the 1-month follow-up visit
* Participation in other studies involving investigational drug(s) within 28 days prior to study entry and/or during study participation

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy women ≥18 and ≤49 years of age.
Enrollment: 306 (Actual)
Dates: Start 2022-08-12 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- United States (12):
  - Alliance for Multispecialty Research, LLC, Newton, Kansas
  - Quality Clinical Research, Inc, Omaha, Nebraska
  - Alliance for Multispecialty Research, LLC, Las Vegas, Nevada
  - Accellacare - Raleigh, Raleigh, North Carolina
  - Accellacare - Wilmington, Wilmington, North Carolina
  - PriMED Clinical Research, Dayton, Ohio
  - PriMed Clinical Research, Dayton, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Alliance for Multispecialty Research, LLC, Knoxville, Tennessee
  - Benchmark Research, Fort Worth, Texas
  - DM Clinical Research - Brookline, Houston, Texas
  - J. Lewis Research, Inc. / Foothill Family Clinic South, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Smith WB, Seger W, Chawana R, Skogeby Z, Silmon de Monerri NC, Feng Y, Gaylord M, Jongihlati B, Beeslaar J, Skinner JM, Bickham K, Anderson AS. A Phase 2b Trial Evaluating the Safety, Tolerability, and Immunogenicity of a 6-Valent Group B Streptococcus Vaccine Administered Concomitantly With Tetanus, Diphtheria, and Acellular Pertussis Vaccine in Healthy Nonpregnant Female Individuals. J Infect Dis. 2025 Jul 11;231(6):e1065-e1074. doi: 10.1093/infdis/jiaf096. PMID 40036340
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C1091005

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy non-pregnant female participants aged 18-49 years, were randomized to receive multivalent group B streptococcus 6-valent polysaccharide conjugate vaccine (GBS6) and tetanus toxoid, diphtheria toxoid, and acellular pertussis vaccine (Tdap), or GBS6 and placebo, or placebo and Tdap.
Pre-assignment Details: A total of 306 participants were enrolled and randomized in the study, of whom 304 were vaccinated.
Groups:
- GBS6 + Tdap: Participants were randomized to receive GBS6 120 microgram (mcg) (0.5 milliliter [mL]) and Tdap (0.5 mL) intramuscularly in the left and right deltoid muscle respectively on Day 1.
- GBS6 + Placebo: Participants were randomized to receive GBS6 120 mcg (0.5 mL) and placebo (0.5 mL, normal saline) intramuscularly in the left and right deltoid muscle respectively on Day 1.
- Placebo + Tdap: Participants were randomized to receive placebo (0.5 mL normal saline) and Tdap (0.5 mL) intramuscularly in the left and right deltoid muscle respectively on Day 1.
Period: Overall Study
Arm/Group | GBS6 + Tdap | GBS6 + Placebo | Placebo + Tdap
Started | 103 | 99 | 104
Vaccinated | 102 | 99 | 103
Completed | 99 | 93 | 98
Not Completed | 4 | 6 | 6
Not completed — Lost to Follow-up | 3 | 5 | 3
Not completed — Withdrawal by Subject | 1 | 1 | 2
Not completed — Other | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety set included all participants who received at least 1 dose of the study interventions and had at least 1 valid post dose safety assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | GBS6 + Tdap | GBS6 + Placebo | Placebo + Tdap | Total
Number analyzed (Participants) | 102 | 99 | 103 | 304
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.4 (8.54) | 34.8 (8.60) | 35.5 (8.59) | 35.3 (8.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 99 | 103 | 304
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 12 | 16 | 36
  Not Hispanic or Latino | 93 | 86 | 86 | 265
  Unknown or Not Reported | 1 | 1 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 0 | 4
  Asian | 3 | 5 | 1 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 18 | 19 | 19 | 56
  White | 80 | 68 | 75 | 223
  More than one race | 0 | 4 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting Local Reactions Within 7 Days After Vaccination
Description: Local reactions (redness, swelling, and pain at the injection site of the left arm) were recorded by participants in e-diary. Erythema/Redness and induration/swelling were measured and recorded in measuring device units (1 measuring device unit=0.5 centimeter [cm]). Grading: Grade 1/mild (greater than [>] 2.0 to 5.0 cm), Grade 2/moderate (>5.0 to 10.0 cm), Grade 3/severe (>10.0 cm) and Grade 4 (necrosis [swelling] or necrosis or exfoliative dermatitis [redness]). Pain at injection site was graded as Grade 1/mild (did not interfere with activity), Grade2/moderate (interfered with activity), Grade 3/severe (prevented daily activity) and Grade 4 (emergency room [ER] visit or hospitalization for severe pain at injection site). Grade 4 were classified by investigator or medically qualified person.
Time Frame: Day 1 (day of vaccination) to Day 7
Population: Safety set included all participants who received at least 1 dose of the study interventions and had at least 1 valid post dose safety assessment. Here, "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | GBS6 + Tdap | GBS6 + Placebo | Placebo + Tdap
Number analyzed (Participants) | 102 | 98 | 103
Percentage of participants
  Pain at injection site: Any | 39.2 [29.7 to 49.4] | 45.9 [35.8 to 56.3] | 33.0 [24.1 to 43.0]
  Pain at injection site: Mild | 27.5 [19.1 to 37.2] | 35.7 [26.3 to 46.0] | 26.2 [18.0 to 35.8]
  Pain at injection site: Moderate | 11.8 [6.2 to 19.6] | 9.2 [4.3 to 16.7] | 6.8 [2.8 to 13.5]
  Pain at injection site: Severe | 0 [0.0 to 3.6] | 1.0 [0.0 to 5.6] | 0 [0.0 to 3.5]
  Pain at injection site: Grade 4 | 0 [0.0 to 3.6] | 0 [0.0 to 3.7] | 0 [0.0 to 3.5]
  Erythema/redness: Any | 7.8 [3.4 to 14.9] | 2.0 [0.2 to 7.2] | 0 [0.0 to 3.5]
  Erythema/redness: Mild | 4.9 [1.6 to 11.1] | 1.0 [0.0 to 5.6] | 0 [0.0 to 3.5]
  Erythema/redness: Moderate | 2.9 [0.6 to 8.4] | 1.0 [0.0 to 5.6] | 0 [0.0 to 3.5]
  Erythema/redness: Severe | 0 [0.0 to 3.6] | 0 [0.0 to 3.7] | 0 [0.0 to 3.5]
  Erythema/redness: Grade 4 | 0 [0.0 to 3.6] | 0 [0.0 to 3.7] | 0 [0.0 to 3.5]
  Induration/swelling: Any | 3.9 [1.1 to 9.7] | 4.1 [1.1 to 10.1] | 1.9 [0.2 to 6.8]
  Induration/swelling: Mild | 1.0 [0.0 to 5.3] | 2.0 [0.2 to 7.2] | 0 [0.0 to 3.5]
  Induration/swelling: Moderate | 2.9 [0.6 to 8.4] | 2.0 [0.2 to 7.2] | 1.9 [0.2 to 6.8]
  Induration/swelling: Severe | 0 [0.0 to 3.6] | 0 [0.0 to 3.7] | 0 [0.0 to 3.5]
  Induration/swelling: Grade 4 | 0 [0.0 to 3.6] | 0 [0.0 to 3.7] | 0 [0.0 to 3.5]

2. Primary Outcome: Percentage of Participants Reporting Systemic Reactions Within 7 Days After Vaccination
Description: Systemic events were recorded in e-diary. Fever: oral temperature greater than or equal to (>=) 38.0 degree Celsius (deg C) and categorized as >=38.0-38.4 deg C, >38.4-38.9 deg C, >38.9-40.0 deg C and >40.0 deg C. Nausea/vomiting was graded as: Grade 1/mild (1-2 times in 24 hours [h]), Grade 2/moderate: (>2 times in 24h), Grade 3/severe (required intravenous hydration) and Grade 4 (ER visit/hospitalization for hypotensive shock). Diarrhea was graded as: Grade 1/mild (2-3 loose stools in 24h), Grade 2/moderate (4-5 loose stools in 24h), Grade 3/severe (6 or more loose stools in 24h) and Grade 4 (ER visit/hospitalization for severe diarrhea). Fatigue/tiredness, headache, chills, muscle pain and joint pain were graded as: Grade 1/mild (did not interfere with activity), Grade 2/moderate (some interference with activity), Grade 3/severe (prevented daily routine activity) and Grade 4 (ER visit/hospitalization). Grade 4 were classified by investigator or medically qualified person.
Time Frame: Day 1 (day of vaccination) to Day 7
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | GBS6 + Tdap | GBS6 + Placebo | Placebo + Tdap
Number analyzed (Participants) | 102 | 99 | 103
Percentage of participants
  Fever: >= 38.0°C | 1.0 [0.0 to 5.3] | 4.0 [1.1 to 10.1] | 2.9 [0.6 to 8.3]
  Fever: 38.0°C to 38.4°C | 0 [0.0 to 3.6] | 2.0 [0.2 to 7.2] | 2.9 [0.6 to 8.3]
  Fever: >38.4°C to 38.9°C | 1.0 [0.0 to 5.3] | 0 [0.0 to 3.7] | 0 [0.0 to 3.5]
  Fever: >38.9°C to 40.0°C | 0 [0.0 to 3.6] | 2.0 [0.2 to 7.2] | 0 [0.0 to 3.5]
  Fever: >40.0°C | 0 [0.0 to 3.6] | 0 [0.0 to 3.7] | 0 [0.0 to 3.5]
  Nausea/vomiting: Any | 14.7 [8.5 to 23.1] | 17.2 [10.4 to 26.3] | 14.6 [8.4 to 22.9]
  Nausea/vomiting: Mild | 7.8 [3.4 to 14.9] | 12.1 [6.5 to 20.4] | 12.6 [6.9 to 20.6]
  Nausea/vomiting: Moderate | 6.9 [2.8 to 13.6] | 5.1 [1.7 to 11.5] | 1.9 [0.2 to 6.8]
  Nausea/vomiting: Severe | 0 [0.0 to 3.6] | 0 [0.0 to 3.7] | 0 [0.0 to 3.5]
  Nausea/vomiting: Grade 4 | 0 [0.0 to 3.6] | 0 [0.0 to 3.7] | 0 [0.0 to 3.5]
  Diarrhea: Any | 19.6 [12.4 to 28.6] | 16.2 [9.2 to 25.2] | 21.4 [13.9 to 30.5]
  Diarrhea: Mild | 15.7 [9.2 to 24.2] | 11.1 [5.7 to 19.2] | 13.6 [7.6 to 21.8]
  Diarrhea: Moderate | 3.9 [1.1 to 9.7] | 4.0 [1.1 to 10.1] | 7.8 [3.4 to 14.7]
  Diarrhea: Severe | 0 [0.0 to 3.6] | 1.0 [0.0 to 5.6] | 0 [0.0 to 3.5]
  Diarrhea: Grade 4 | 0 [0.0 to 3.6] | 0 [0.0 to 3.7] | 0 [0.0 to 3.5]
  Headache: Any | 35.3 [26.1 to 45.4] | 48.5 [38.3 to 58.7] | 38.8 [29.4 to 48.9]
  Headache: Mild | 23.5 [15.7 to 33.0] | 34.3 [25.1 to 44.6] | 26.2 [18.0 to 35.8]
  Headache: Moderate | 10.8 [5.5 to 18.5] | 13.1 [7.2 to 21.4] | 12.6 [6.9 to 20.6]
  Headache: Severe | 1.0 [0.0 to 5.3] | 1.0 [0.0 to 5.5] | 0 [0.0 to 3.5]
  Headache: Grade 4 | 0 [0.0 to 3.6] | 0 [0.0 to 3.7] | 0 [0.0 to 3.5]
  Fatigue/tiredness: Any | 51.0 [40.9 to 61.0] | 50.5 [40.7 to 61.3] | 46.6 [36.7 to 56.7]
  Fatigue/tiredness: Mild | 29.4 [20.8 to 39.3] | 21.2 [13.8 to 30.9] | 19.4 [12.3 to 28.4]
  Fatigue/tiredness: Moderate | 20.6 [13.2 to 29.7] | 24.2 [16.4 to 34.2] | 26.2 [18.0 to 35.8]
  Fatigue/tiredness: Severe | 1.0 [0.0 to 5.3] | 5.1 [1.7 to 11.5] | 1.0 [0.0 to 5.3]
  Fatigue/tiredness: Grade 4 | 0 [0.0 to 3.6] | 0 [0.0 to 3.7] | 0 [0.0 to 3.5]
  Muscle pain: Any | 30.4 [21.7 to 40.3] | 24.2 [16.4 to 34.2] | 26.2 [18.0 to 35.8]
  Muscle pain: Mild | 14.7 [8.5 to 23.1] | 13.1 [7.3 to 21.6] | 14.6 [8.4 to 22.9]
  Muscle pain: Moderate | 15.7 [9.2 to 24.2] | 10.1 [5.0 to 18.0] | 11.7 [6.2 to 19.5]
  Muscle pain: Severe | 0 [0.0 to 3.6] | 1.0 [0.0 to 5.6] | 0 [0.0 to 3.5]
  Muscle pain: Grade 4 | 0 [0.0 to 3.6] | 0 [0.0 to 3.7] | 0 [0.0 to 3.5]
  Joint pain: Any | 17.6 [10.8 to 26.4] | 15.2 [8.8 to 24.0] | 12.6 [6.9 to 20.6]
  Joint pain: Mild | 9.8 [4.8 to 17.3] | 10.1 [5.0 to 18.0] | 5.8 [2.2 to 12.2]
  Joint pain: Moderate | 7.8 [3.4 to 14.9] | 3.0 [0.6 to 8.7] | 6.8 [2.8 to 13.5]
  Joint pain: Severe | 0 [0.0 to 3.6] | 2.0 [0.2 to 7.2] | 0 [0.0 to 3.5]
  Joint pain: Grade 4 | 0 [0.0 to 3.6] | 0 [0.0 to 3.7] | 0 [0.0 to 3.5]

3. Primary Outcome: Percentage of Participants Reporting Adverse Events (AEs) Through 1 Month After Vaccination
Description: An AE was any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. In this outcome measure results excluded data for local reactions and systemic events.
Time Frame: Day 1 (day of vaccination) through 1 Month post-vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | GBS6 + Tdap | GBS6 + Placebo | Placebo + Tdap
Number analyzed (Participants) | 102 | 99 | 103
Percentage of participants | 5.9 [2.2 to 12.4] | 8.1 [3.6 to 15.3] | 3.9 [1.1 to 9.6]

4. Primary Outcome: Percentage of Participants Reporting Medically Attended Adverse Events (MAEs) and Serious Adverse Events (SAEs) Through 6 Months After Vaccination
Description: A MAE was defined as a non-serious AE that resulted in an evaluation at a medical facility. A SAE was defined as any untoward medical occurrence at any dose that resulted in any of the following outcomes: death; life-threatening (immediate risk of death); required inpatient hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); congenital anomaly/birth defect; or that was considered as an important medical event.
Time Frame: Day 1 (day of vaccination) through 6 Months post-vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | GBS6 + Tdap | GBS6 + Placebo | Placebo + Tdap
Number analyzed (Participants) | 102 | 99 | 103
Percentage of participants
  MAEs | 4.9 [1.6 to 11.1] | 4.0 [1.1 to 10.0] | 6.8 [2.8 to 13.5]
  SAEs | 0 [0.0 to 3.6] | 0 [0.0 to 3.7] | 1.0 [0.0 to 5.3]

5. Primary Outcome: Percentage of Participants Achieving Anti-tetanus Toxoid (Anti-TTd) and Anti-diphtheria Toxoid (Anti-DTd) Antibody Concentration >=0.1 IU/mL at 1 Month After Vaccination: GBS6 + Tdap and Placebo + Tdap Groups
Description: IU/mL stands for international units per milliliter.
Time Frame: 1 Month after Vaccination (Day 1, day of vaccination)
Population: Evaluable immunogenicity population included all participants who were eligible, received all doses of the investigational products to which they were randomized, had blood drawn for assay testing within the specified time frame for 1 month after vaccination, had at least 1 valid and determinate assay result at the 1-month postvaccination visit, and had no major protocol violations.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | GBS6 + Tdap | Placebo + Tdap
Number analyzed (Participants) | 99 | 101
Percentage of participants
  Anti-TTd | 100.0 [96.3 to 100.0] | 100.0 [96.4 to 100.0]
  Anti-DTd | 100.0 [96.3 to 100.0] | 100.0 [96.4 to 100.0]
Statistical Analysis 1: Comparison: GBS6 + Tdap vs Placebo + Tdap; Test type: Other; Risk difference = 0.0, 95% CI [-3.8 to 3.7]

6. Primary Outcome: Geometric Mean Concentration (GMC) of Anti-Pertussis Toxin (PT), Anti-Filamentous Hemagglutinin (FHA), and Anti-Pertactin (PRN) Antibodies; GMR of Anti-PT, Anti-FHA, and Anti-PRN for GBS6 + Tdap to Placebo + Tdap at 1 Month After Vaccination
Description: GMCs of anti-PT, anti-FHA, and anti-PRN was reported as descriptive data for the GBS6 +Tdap and placebo + Tdap groups, along with associated 2-sided 95% confidence interval. GMR for anti-PT, anti-FHA and anti-PRN antibodies were estimated from the GBS6 + Tdap group to the placebo + Tdap group and reported as statistical data.
Time Frame: 1 Month after Vaccination (Day 1, day of vaccination)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Endotoxin units per milliliter (EU/mL)
Arm/Group | GBS6 + Tdap | Placebo + Tdap
Number analyzed (Participants) | 99 | 101
Endotoxin units per milliliter (EU/mL)
  GMC of Anti-PT antibodies | 17.975 [14.519 to 22.254] | 32.916 [26.641 to 40.668]
  GMC of Anti-FHA antibodies | 108.377 [93.479 to 125.650] | 191.140 [161.964 to 225.571]
  GMC of Anti-PRN antibodies | 158.887 [132.346 to 190.751] | 270.294 [222.691 to 328.072]
Statistical Analysis 1: Comparison: GBS6 + Tdap vs Placebo + Tdap; GMR for Anti-PT Antibody: GMR for GBS6 + Tdap/Placebo + Tdap was calculated by back transforming the mean difference between the 2 measures on the logarithmic scale; Test type: Other; GMR = 0.546, 95% CI 2-sided [0.405 to 0.736]
Statistical Analysis 2: Comparison: GBS6 + Tdap vs Placebo + Tdap; GMR for Anti-FHA Antibody: GMR for GBS6 + Tdap/Placebo + Tdap was calculated by back transforming the mean difference between the 2 measures on the logarithmic scale; Test type: Other; GMR = 0.567, 95% CI 2-sided [0.455 to 0.707]
Statistical Analysis 3: Comparison: GBS6 + Tdap vs Placebo + Tdap; GMR for Anti-PRN Antibody: GMR for GBS6 + Tdap/Placebo + Tdap was calculated by back transforming the mean difference between the 2 measures on the logarithmic scale; Test type: Other; GMR = 0.588, 95% CI 2-sided [0.451 to 0.766]

7. Primary Outcome: GMC of GBS Capsular Polysaccharide (CPS) Serotype-Specific Immunoglobulin G (IgG) Antibodies; GMR of GBS CPS Serotype-specific IgG Antibodies for GBS6 + Tdap to Placebo + Tdap at 1 Month After Vaccination
Description: GBS CPS serotype-specific IgG GMCs (Ia, Ib, II, III, IV, V) were reported as descriptive data for the GBS6+Tdap and GBS6+placebo groups, along with associated 2-sided 95% confidence interval. GMR of GBS CPS serotype-specific IgG antibodies were estimated from the GBS6 + Tdap group to the placebo + Tdap group and reported as statistical data.
Time Frame: 1 Month after Vaccination (Day 1, day of vaccination)
Population: Evaluable immunogenicity population evaluated. Here, "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure. Here, "Number analyzed" signifies number of participants with valid and determinate assay results for the serotype at the specified time point.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | GBS6 + Tdap | GBS6 + Placebo
Number analyzed (Participants) | 99 | 94
mcg/mL
  Ia: number analyzed (Participants) | 98 | 94
  Ia | 13.015 [7.095 to 23.874] | 14.616 [7.965 to 26.821]
  Ib | 2.421 [1.322 to 4.431] | 2.106 [1.037 to 4.278]
  II | 63.656 [40.279 to 100.600] | 61.709 [39.961 to 95.291]
  III: number analyzed (Participants) | 98 | 93
  III | 3.521 [2.107 to 5.885] | 5.547 [3.239 to 9.500]
  IV: number analyzed (Participants) | 97 | 94
  IV | 6.065 [4.097 to 8.980] | 4.115 [2.746 to 6.167]
  V | 1.307 [0.722 to 2.363] | 2.337 [1.209 to 4.517]
Statistical Analysis 1: Comparison: GBS6 + Tdap vs GBS6 + Placebo; GMR for serotype Ia: GMR for GBS6 + GBS6/Placebo + Tdap was calculated by back transforming the mean difference between the 2 measures on the logarithmic scale; Test type: Other; GMR = 0.890, 95% CI 2-sided [0.380 to 2.089]
Statistical Analysis 2: Comparison: GBS6 + Tdap vs GBS6 + Placebo; GMR for serotype Ib: GMR for GBS6 + GBS6/Placebo + Tdap was calculated by back transforming the mean difference between the 2 measures on the logarithmic scale; Test type: Other; GMR = 1.149, 95% CI 2-sided [0.455 to 2.901]
Statistical Analysis 3: Comparison: GBS6 + Tdap vs GBS6 + Placebo; GMR for serotype II: GMR for GBS6 + GBS6/Placebo + Tdap was calculated by back transforming the mean difference between the 2 measures on the logarithmic scale; Test type: Other; GMR = 1.032, 95% CI [0.551 to 1.931]
Statistical Analysis 4: Comparison: GBS6 + Tdap vs GBS6 + Placebo; GMR for serotype III: GMR for GBS6 + GBS6/Placebo + Tdap was calculated by back transforming the mean difference between the 2 measures on the logarithmic scale; Test type: Other; GMR = 0.635, 95% CI 2-sided [0.303 to 1.329]
Statistical Analysis 5: Comparison: GBS6 + Tdap vs GBS6 + Placebo; GMR for serotype IV: GMR for GBS6 + GBS6/Placebo + Tdap was calculated by back transforming the mean difference between the 2 measures on the logarithmic scale; Test type: Other; GMR = 1.474, 95% CI 2-sided [0.842 to 2.580]
Statistical Analysis 6: Comparison: GBS6 + Tdap vs GBS6 + Placebo; GMR for serotype V: GMR for GBS6 + GBS6/Placebo + Tdap was calculated by back transforming the mean difference between the 2 measures on the logarithmic scale; Test type: Other; GMR = 0.559, 95% CI 2-sided [0.232 to 1.349]

ADVERSE EVENTS:
Time Frame: Local reaction and systemic events (systematic assessment): up to 7 days post-vaccination; All-cause mortality, SAEs, MAEs (non-systematic assessment): up to 6 months post-vaccination; Other AEs (non-systematic assessment): up to 1-month post-vaccination [vaccination was on Day 1]
Description: All participants who receive at least 1 dose of the investigational products and have at least 1 valid post dose assessment.
Arm/Group | GBS6 + Tdap | GBS6 + Placebo | Placebo + Tdap
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/99 | 0/103
Serious Adverse Events (participants affected / at risk) | 0/102 | 0/99 | 1/103
Other Adverse Events (participants affected / at risk) | 81/102 | 71/99 | 79/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GBS6 + Tdap (N=102) | GBS6 + Placebo (N=99) | Placebo + Tdap (N=103)
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GBS6 + Tdap (N=102) | GBS6 + Placebo (N=99) | Placebo + Tdap (N=103)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 0 | 0 | 1
Autoimmune thyroiditis (Endocrine disorders) | 0 | 1 | 0
Tooth impacted (Gastrointestinal disorders) | 1 | 0 | 0
Axillary pain (General disorders) | 1 | 0 | 0
Bacterial vaginosis (Infections and infestations) | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 2 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 1
Post procedural infection (Infections and infestations) | 1 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0
Abnormal weight gain (Metabolism and nutrition disorders) | 1 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 0
Nerve compression (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Diarrhoea (DIARRHEA) (Gastrointestinal disorders) | 20 | 16 | 22
Vomiting (NAUSEA/VOMITING) (Gastrointestinal disorders) | 15 | 17 | 15
Fatigue (FATIGUE) (General disorders) | 52 | 50 | 48
Injection site erythema (REDNESS) (General disorders) | 8 | 2 | 0
Injection site pain (PAIN) (General disorders) | 40 | 45 | 34
Injection site swelling (SWELLING) (General disorders) | 4 | 4 | 2
Pyrexia (FEVER) (General disorders) | 1 | 4 | 3
Arthralgia (JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 18 | 15 | 13
Myalgia (MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 31 | 24 | 27
Headache (HEADACHE) (Nervous system disorders) | 36 | 48 | 40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-10-04): https://cdn.clinicaltrials.gov/large-docs/86/NCT04766086/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-14): https://cdn.clinicaltrials.gov/large-docs/86/NCT04766086/SAP_001.pdf